CLINICAL TRIAL: NCT07308275
Title: Longitudinal Evaluation of Direct Neurotization Technique in Breast Reconstruction With Fully Autologous Components: An Assessment of BREAST-Q Sensation Module, Cutaneous Pressure Threshold, Neuregulin 1 (NRG1) Expression, Nerve Fiber Cross-sectional Area, Intraepidermal Nerve Fiber Density (IENFD), and Breast Morphometry
Brief Title: Longitudinal Evaluation of Direct Neurotization Technique in Breast Reconstruction With Fully Autologous Components
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Mohamad Rachadian Ramadan, dr. Mohamad Rachadian Ramadan, B.Med.Sc, Sp.B.P.R.E, Subsp.M.O.(K), MRBS, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDINEUROTISASI
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Reconstruction After Mastectomy; Neurotization; Mastectomy and Breast Reconstruction; Peripheral Nerve Regeneration; Sensory Function; Quality of Life (QOL)
Keywords: breast neurotization; mastectomy; breast sensory; quality of life
MeSH Terms: interventions — Nerve Transfer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Neurotized Group (Active Comparator): Participants assigned to this arm are women undergoing mastectomy who are eligible for standard autologous breast reconstruction without neurotization.
  Interventions: Procedure: Autologous Breast Reconstruction without Neurotization
- Neurotized Group (Experimental): Participants assigned to this arm are women undergoing mastectomy who are eligible for autologous breast reconstruction with planned direct neurotization using fully autologous components.
  Interventions: Procedure: Autologous Breast Reconstruction With Direct Neurotization

INTERVENTIONS:
Procedure: Autologous Breast Reconstruction With Direct Neurotization — The direct neurotization using fully autologous components procedures include:
  1. Direct neurotization is carried out using fully autologous components, involving coaptation of the recipient nerve to an autologous nerve graft placed within the flap to facilitate reinnervation.
  2. Surgical breast reconstruction is then completed using patient's own tissue
  Arms: Neurotized Group
Procedure: Autologous Breast Reconstruction without Neurotization — Breast reconstruction is performed using autologous tissue without nerve coaptation or neurotization, according to standard surgical practice.
  Arms: Non-Neurotized Group

SUMMARY:
This clinical trial aims to evaluate whether direct neurotization using fully autologous components during autologous breast reconstruction improves postoperative breast sensation and sensory-related quality of life in women undergoing unilateral mastectomy. Direct neurotization involves coapting the recipient intercostal nerve to an autologous nerve graft placed within the flap to facilitate reinnervation.

The study's primary questions are:

1. Does direct neurotization using fully autologous nerve grafts improve cutaneous sensory recovery, as assessed by Semmes-Weinstein monofilament thresholds measured at standardized breast locations?
2. Does neurotization enhance patient-reported sensory outcomes and quality of life, as assessed by the BREAST-Q Sensation Module?

As secondary objectives, the study will assess whether biological predictors of nerve regeneration correlate with sensory outcomes. These include:

1. Neuregulin-1 (NRG1) expression in flap tissue biopsy;
2. Cross-sectional area of the recipient nerve fibres;
3. Breast morphometry measured at baseline and follow-up;
4. Intraepidermal nerve fibre density (IENFD) on skin biopsy.

Participants will be randomly assigned to receive either:

1. Neurotized autologous breast reconstruction using fully autologous graft components, or
2. Standard (non-neurotized) autologous breast reconstruction.

The study will compare these groups to determine whether neurotization accelerates or enhances the return of breast sensation over a 6-month follow-up period, with evaluations at 1 month, 3 months, and 6 months after surgery.

Participants will undergo:

1. Autologous breast reconstruction with or without direct neurotization as part of their planned cancer surgery.
2. Sensory testing using Semmes-Weinstein monofilaments at baseline, 1, 3, and 6 months.
3. Completion of BREAST-Q questionnaires evaluating breast sensation, symptoms, and quality of life at each follow-up visit.

3. Intraoperative tissue sampling for NRG1 analysis and nerve morphometry. 4. Skin biopsy (if applicable) to assess intraepidermal nerve fibre density. 5. Breast morphometry assessment using a breast morphometry measurement software tool.

This study seeks to provide high-quality evidence on the effectiveness of direct neurotization using fully autologous components in restoring breast sensation and to explore biological predictors that may influence sensory recovery after autologous breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Patients with unilateral breast cancer who have undergone or will undergo unilateral mastectomy.
* Patients undergoing breast reconstruction.
* Patients with unilateral breast cancer regardless of adjuvant therapy status (receiving radiotherapy and/or chemotherapy or receiving no adjuvant therapy).
* Willing to comply with all scheduled examinations and tissue sampling procedures.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* History of peripheral neuropathy (e.g., diabetes mellitus with neuropathic complications).
* Bilateral mastectomy.
* Presence of skin or soft-tissue conditions of the breast that may interfere with sensory assessment.
* Active smokers (use of tobacco, vape, or other nicotine products within 14 days prior to neurotization).
* Refusal or inability to attend follow-up evaluations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Breast Sensation assessed by using Semmes-Weinstein Monofilament testing | 1, 3 and 6 months after Neurotization
  SWM thresholds at nine standardized points on the reconstructed breast will be measured using calibrated monofilaments, categorized into levels of normal touch, diminished light touch, diminished protective sensation, loss of protective sensation, and deep pressure only.
Patient's Quality of Life assessed by using BREAST-Q® Sensation Module | 1, 3 and 6 months after Neurotization
  The patient reported outcomes will be recorded in BREAST-Q® Sensation Module to capture the sensation, breast symptoms, and quality of life impact of sensation loss.

SECONDARY OUTCOMES:
Neuregulin 1 Expression | During procedure and 6 months after surgery
  NRG1 expression quantified by ELISA from flap tissue
Nerve Cross-sectional Area | Measured during neurotization procedure
  Nerve cross-sectional area measured via histomorphometry/histopathology using the recipient nerve of the direct neurotization method
Breast Morphometry | Before surgery and 1, 3, 6 months after surgery
  Breast morphometry assessed using a validated AR/3D application
Intraepidermal Nerve Fibre Density (IENFD) | During procedure and 6 months after surgery
  IENFD quantified by counting PGP9.5-positive intraepidermal fibers per mm of epidermal length. Flap skin tissue samples will be taken using 3 mm punch biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- dr. Ciptomangunkusumo National Hospital - Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding participant confidentiality and the potential risk of re-identification in a small surgical trial with detailed clinical and biomarker data.

REFERENCES:
- [Background] Bubberman JM, Brandts L, van Kuijk SMJ, van der Hulst RRWJ, Tuinder SMH. The efficacy of sensory nerve coaptation in DIEP flap breast reconstruction - Preliminary results of a double-blind randomized controlled trial. Breast. 2024 Apr;74:103691. doi: 10.1016/j.breast.2024.103691. Epub 2024 Feb 9. PMID 38401421
- [Background] Timar B, Popescu S, Timar R, Baderca F, Duica B, Vlad M, Levai C, Balinisteanu B, Simu M. The usefulness of quantifying intraepidermal nerve fibers density in the diagnostic of diabetic peripheral neuropathy: a cross-sectional study. Diabetol Metab Syndr. 2016 Apr 11;8:31. doi: 10.1186/s13098-016-0146-4. eCollection 2016. PMID 27069510
- [Background] Samolis A, Troupis T, Politis C, Pantazis N, Triantafyllou G, Tsakotos G, Tegos T, Lazaridis N, Natsis K, Piagkou M. Intraepidermal Nerve Fiber Density as an Indicator of Neuropathy Predisposition: A Systematic Review with Meta-Analysis. Diagnostics (Basel). 2025 May 23;15(11):1311. doi: 10.3390/diagnostics15111311. PMID 40506883
- [Background] La Padula S, Pensato R, D'Andrea F, de Gregorio L, Errico C, Rega U, Canta L, Pizza C, Roccaro G, Billon R, Dibra E, Meningaud JP, Hersant B. Assessment of Patient Satisfaction Using a New Augmented Reality Simulation Software for Breast Augmentation: A Prospective Study. J Clin Med. 2022 Jun 16;11(12):3464. doi: 10.3390/jcm11123464. PMID 35743534
- [Background] Song S, Parmeshwar N, Steiner G, Kim EA. Morphometric Analysis of Gender-affirming Breast Augmentation. Plast Reconstr Surg Glob Open. 2022 Nov 29;10(11):e4691. doi: 10.1097/GOX.0000000000004691. eCollection 2022 Nov. PMID 36467119
- [Background] Bin JM, Suminaite D, Benito-Kwiecinski SK, Kegel L, Rubio-Brotons M, Early JJ, Soong D, Livesey MR, Poole RJ, Lyons DA. Importin 13-dependent axon diameter growth regulates conduction speeds along myelinated CNS axons. Nat Commun. 2024 Feb 27;15(1):1790. doi: 10.1038/s41467-024-45908-6. PMID 38413580
- [Background] Clark IA, Mohammadi S, Callaghan MF, Maguire EA. Conduction velocity along a key white matter tract is associated with autobiographical memory recall ability. Elife. 2022 Sep 27;11:e79303. doi: 10.7554/eLife.79303. PMID 36166372
- [Background] Fricker FR, Lago N, Balarajah S, Tsantoulas C, Tanna S, Zhu N, Fageiry SK, Jenkins M, Garratt AN, Birchmeier C, Bennett DL. Axonally derived neuregulin-1 is required for remyelination and regeneration after nerve injury in adulthood. J Neurosci. 2011 Mar 2;31(9):3225-33. doi: 10.1523/JNEUROSCI.2568-10.2011. PMID 21368034
- [Background] Stassart RM, Fledrich R, Velanac V, Brinkmann BG, Schwab MH, Meijer D, Sereda MW, Nave KA. A role for Schwann cell-derived neuregulin-1 in remyelination. Nat Neurosci. 2013 Jan;16(1):48-54. doi: 10.1038/nn.3281. Epub 2012 Dec 9. PMID 23222914
- [Background] Dellon ES, Crone S, Mouery R, Dellon AL. Comparison of the Semmes-Weinstein monofilaments with the Pressure-Specifying Sensory Device. Restor Neurol Neurosci. 1993 Jan 1;5(5):323-6. doi: 10.3233/RNN-1993-55602. PMID 21551718
- [Background] Voineskos SH, Klassen AF, Cano SJ, Pusic AL, Gibbons CJ. Giving Meaning to Differences in BREAST-Q Scores: Minimal Important Difference for Breast Reconstruction Patients. Plast Reconstr Surg. 2020 Jan;145(1):11e-20e. doi: 10.1097/PRS.0000000000006317. PMID 31577663
- [Background] Gallo L, Chu JJ, Shamsunder MG, Hatchell A, Patel AR, Godwin K, Hernandez M, Pusic AL, Nelson JA, Voineskos SH. Best Practices for BREAST-Q Research: A Systematic Review of Study Methodology. Plast Reconstr Surg. 2022 Sep 1;150(3):526e-535e. doi: 10.1097/PRS.0000000000009401. Epub 2022 Jun 24. PMID 35749737
- [Background] Ramadan MR, Rifai DA, Atmodiwirjo P, Panigoro SS, Mukarramah DA, Sobri FB, Jurisman A, Djohan R. Indonesian Translation and Cultural Adaptation of the BREAST-Q Reconstruction Module. Plast Reconstr Surg Glob Open. 2025 Apr 21;13(4):e6705. doi: 10.1097/GOX.0000000000006705. eCollection 2025 Apr. PMID 40264905
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Shiah E, Laikhter E, Comer CD, Manstein SM, Bustos VP, Bain PA, Lee BT, Lin SJ. Neurotization in Innervated Breast Reconstruction: A Systematic Review of Techniques and Outcomes. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):2890-2913. doi: 10.1016/j.bjps.2022.06.006. Epub 2022 Jun 17. PMID 35872020
- [Background] Tecce MG, Desai AA, Christopher A, Cunning J, Rios-Diaz AJ, Morris MP, et al. 6. Breast Flap Neurotization After Autologous Free Flap Breast Reconstruction: A Prospective Trial. In: PRS Global Open [Internet]. 2022. Available from: http://journals.lww.com/prsgo
- [Background] Shyu S, Chang TN, Lu JC, Chen CF, Cheong DC, Kao SW, Kuo WL, Huang JJ. Breast neurotization along with breast reconstruction after nipple sparing mastectomy enhances quality of life and reduces denervation symptoms in patient-reported outcome: a prospective cohort study. Int J Surg. 2025 May 1;111(5):3235-3247. doi: 10.1097/JS9.0000000000002331. PMID 40072353
- [Background] Jagasia PM, Bagdady K, Jordan SW, Howard MA, Fracol ME. Meta-analysis of Objective Sensory Outcomes From 764 Breasts Shows Superior Sensation of Autologous Reconstruction With Neurotization. Plast Reconstr Surg Glob Open. 2025 May 6;13(5):e6751. doi: 10.1097/GOX.0000000000006751. eCollection 2025 May. PMID 40330161